CLINICAL TRIAL: NCT05127798
Title: Real World Evidence of First Line Treatment With Intensive Chemotherapy in Adult Patients With Acute Myeloid Leukemia From 18 to 70 Years Old
Brief Title: RWE of 1st Line Treatment in Adults With AML From 18 to 70 Years Old.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grupo Argentino de Tratamiento de la Leucemia Aguda (Other)
Responsible Party: Sponsor
Other Study IDs: GATLA 10-LMA-20
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Acute Myeloid Leukemia, Adult
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult from 18 to 70 years old AML in first line: Patients >/= 18 years old with recent diagnosis of AML who receive treatment with intensive chemotherapy according to our local guidelines.
  Interventions: Other: Evaluation of first line treatment with intensive treatment outcome in adult patients with AML.

INTERVENTIONS:
Other: Evaluation of first line treatment with intensive treatment outcome in adult patients with AML. — Evaluation of first line treatment with intensive treatment outcome (or event free survival and overall survival and toxicity) in adult patients between 18 and 70 years old with AML.

SUMMARY:
This is a multicenter, observational real world clinical trial with prospective follow up that will evaluate the treatment outcome of Acute Myeloid Leukemia (AML) patients in the first line with intensive chemotherapy based regimens in Argentina.

DETAILED DESCRIPTION:
The purpose of this trial is to gather real world evidence of the characteristics of AML patients in Argentina who receive intensive chemotherapy based treatment in first line following our national guidelines. The study primary endpoint is to evaluate event free survival (EFS) and overall survival (OS) of patients diagnosed with AML and treated in first line with intensive chemotherapy combined with different consolidation modalities depending on risk category. Secondary endpoints are to evaluate EFS and OS according to: cytogenetic and molecular classification, measurable residual disease (MRD) (by flow cytometry) post induction. Assess treatment-related mortality and limitations in completing treatment due to toxicity. Evaluate the role of allogeneic stem cell transplantation in terms of EFS in intermediate and adverse risk patients.

Every AML patient diagnosed in our institutions will follow our guidelines with respect to diagnosis procedures. Risk category will depend on molecular and cytogenetic features according to European Leukemia net 2017 risk stratification.

All patients will receive induction with 7+3 scheme; if CR is not met induction will be followed by a reinduction with FLAG-IDA. According to post induction remission status and risk assessment, consolidation will consist of three courses of cytarabine (2g/m2) + daunorubicin (60mg/m2) for low risk group; or consolidation with cytarabine (2g/m2) + daunorubicin (60mg/m2) followed by allogeneic stem cell transplantation for intermediate and adverse risk groups.

Patients harboring Flt3 mutation will add midostaurin during induction and consolidations: midostaurin 50 mg orally every 12 hours on days 8-21 of each 28-day cycle.

In the cases of Coring Binding Factor AML and NPM1 mutated AML, molecular MRD assessment will be done at the end of consolidations by RQ-PCR and thereafter a follow-up RQ-PCR evaluation every 3 months during the first two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.
* Patients with AML (de novo or secondary to MDS or previous treatment) who meet the diagnostic criteria according to WHO 2016 classification.
* Signature of the form consent for participation in the study.

Exclusion Criteria:

* Men and women, <18 or >70 years of age.
* Patients with chronic myeloid leukemia blast crisis or transformation to acute leukemia of other myeloproliferative syndromes.
* Patients with relapsed AML.
* Acute promyelocytic leukemia t(15; 17) or variants.
* Absence of written informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status ≥ 3 that is not due to the disease that motivates the treatment (AML).
* Transplant Comorbidity Index (HCT-CI) >3.
* Left ventricular ejection fraction < 40% by echocardiogram (Simpsom).
* Bilirubin, alkaline phosphatase or alanine aminotransferase > 3 times the upper normal limit not due to AML.
* Serum creatinine ≥ 2.5 mg/dL not due to AML.
* Positive pregnancy test or absence of effective methods of contraception in women of childbearing age.
* Presence of active neoplasia other than AML whose treatment is more urgent at the discretion of the treating physicians.
* Presence of serious psychiatric illness.
* Known history of infection with human immunodeficiency virus (HIV). Active uncontrolled Hepatitis C or Active uncontrolled Hepatitis B.
* Any other condition, such as age or associated pathology that contraindicates treatment with intensive chemotherapy, especially with anthracyclines. Any patient who does not meet the inclusion and exclusion criteria for treatment with intensive chemotherapy may be evaluated on an individual basis if it is considered that they could still benefit from this treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients between 18 and 70 years old with AML in first line treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Overall Survival of patients diagnosed with primary or secondary AML between 18 and 70 years of age treated in first line with intensive chemotherapy regimens and risk-adapted consolidation. | 36 months
  Evaluate overall survival of patients diagnosed with AML and treated in first line with intensive chemotherapy combined with different consolidation modalities depending on risk category
Evaluate the Event Free Survival of patients diagnosed with primary or secondary AML between 18 and 70 years of age treated in first line with intensive chemotherapy regimens and risk-adapted consolidation. | 36 months
  Evaluate the Event Free Survival of patients diagnosed with AML and treated in first line with intensive chemotherapy combined with different consolidation modalities depending on risk category.

SECONDARY OUTCOMES:
Evaluate the Complete Remission Rate with negative measurable residual disease (MRD) determined by CMF at the end of induction treatment. | 36 months
Evaluate the toxicity of the scheme measured by type, frequency, severity and relation to treatment of adverse events. | 36 months
Evaluate treatment-related mortality (within 30 days of admission). | Within 30 days of admission
Evaluate the role of measurable residual disease (MRD) in terms of EFS prior to each consolidation. | 36 months
Evaluate the role of allogeneic stem cell transplantation in terms of EFS in intermediate and adverse risk patients. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose Mela Osorio, Dr., Principal Investigator — Grupo Argentino de Tratamiento de la Leucemia Aguda; Hernan Dick, Dr., Principal Investigator — Grupo Argentino de Tratamiento de la Leucemia Aguda; Isolda Fernandez, Dr., Study Chair — Grupo Argentino de Tratamiento de la Leucemia Aguda
Locations (2):
- Argentina (2):
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - FUNDALEU, CABA

IPD SHARING:
Plan to Share IPD: Yes
Share study protocol
Supporting Information: Study Protocol
Time Frame: The data is available since June 2021, and will remain available until the end of the clinical trial.